CLINICAL TRIAL: NCT00589316
Title: Hematopoietic Bone Marrow Transplantation for Patients With High-risk Acute Myeloid Leukemia (AML), Acute Lymphoblastic Leukemia (ALL), or Myelodysplastic Syndrome (MDS) Using Related HLA-Mismatched Donors: A Trial Using Radiolabeled Anti-CD45 Antibody Combined With Immunosuppression Before and After Transplantation
Brief Title: Iodine I 131 Monoclonal Antibody BC8, Fludarabine Phosphate, Cyclophosphamide, Total-Body Irradiation and Donor Bone Marrow Transplant in Treating Patients With Advanced Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia, or High-Risk Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to loss of funding
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Johnnie Orozco, Associate Professor, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2186.00; NCI-2010-00404 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2186.00p; 2186.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA044991 (NIH); RG1707019 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2008-01-03; First posted 2008-01-09 (Estimated); Results first posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; CD45-Positive Neoplastic Cells Present; Chronic Myelomonocytic Leukemia; Previously Treated Myelodysplastic Syndrome; Refractory Anemia With Excess Blasts; Refractory Anemia With Ring Sideroblasts; Refractory Cytopenia With Multilineage Dysplasia; Refractory Cytopenia With Multilineage Dysplasia and Ring Sideroblasts
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Anemia, Refractory, with Excess of Blasts | interventions — Cyclophosphamide; fludarabine phosphate; Iodine-131; Mycophenolic Acid; Tacrolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (chemo, TBI, transplant, immunosuppression) (Experimental): RADIOIMMUNOTHERAPY: Patients receive therapeutic iodine I 131 monoclonal antibody BC8 via central line on day -14.
  NONMYELOABLATIVE CONDITIONING: Patients receive FLU IV over 30 minutes on days -6 to -2 and CY IV over 1 hour on days -6 and -5. Patients undergo TBI on day -1.
  TRANSPLANTATION: Patients undergo allogeneic bone marrow transplantation on day 0.
  POST-TRANSPLATATION IMMUNOSUPPRESSION: Patients receive CY IV over 1-2 hours on day 3, MMF IV or PO TID on days 4 to 35, and tacrolimus IV over 1-2 hours or PO on days 4 to 180 with taper on day 84.
  Interventions: Procedure: Allogeneic Bone Marrow Transplantation; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Radiation: Iodine I 131 Monoclonal Antibody BC8; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Drug: Tacrolimus; Radiation: Total-Body Irradiation

INTERVENTIONS:
Procedure: Allogeneic Bone Marrow Transplantation — Given via central line
  Other Names: Allo BMT; Allogeneic BMT
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Radiation: Iodine I 131 Monoclonal Antibody BC8 — Given IV (dosimetry dose) or via central line (therapeutic dose)
  Other Names: I 131 MOAB BC8; I 131 Monoclonal Antibody BC8; iodine I 131 MOAB BC8; Iomab-B; MOAB BC8, iodine I 131; monoclonal antibody BC8, iodine I 131
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mycophenolate Mofetil — Given IV or PO
  Other Names: Cellcept; MMF
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation

SUMMARY:
This phase I trial studies the side effects and best dose of iodine I 131monoclonal antibody BC8 when given together with fludarabine phosphate, cyclophosphamide, total-body irradiation, and donor bone marrow transplant, and to see how well they work in treating patients with acute myeloid leukemia or acute lymphoblastic leukemia that has spread to nearby or other places in the body (advanced), or high-risk myelodysplastic syndrome. Giving chemotherapy drugs, such as fludarabine phosphate and cyclophosphamide, and total-body irradiation before a donor bone marrow transplant helps stop the growth of cancer or abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. Also, radiolabeled monoclonal antibodies, such as iodine I 131 monoclonal antibody BC8, can find cancer cells and carry cancer-killing substances to them without harming normal cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclophosphamide together with mycophenolate mofetil and tacrolimus after the transplant may stop this from happening. Giving a radiolabeled monoclonal antibody together with donor stem cell transplant, fludarabine phosphate, cyclophosphamide, mycophenolate mofetil, and tacrolimus may be an effective treatment for advanced acute myeloid leukemia, acute lymphoblastic leukemia, or myelodysplastic syndromes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose of radiation delivered via 131 I-BC8 antibody (iodine I 131 monoclonal antibody BC8) when combined with pre- and post-transplant cyclophosphamide (CY), fludarabine phosphate (FLU), 2 Gy total-body irradiation (TBI), tacrolimus, mycophenolate mofetil (MMF), and a haploidentical allogeneic hematopoietic marrow transplant in patients who have advanced acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), or high risk myelodysplastic syndromes (MDS).

II. To estimate rates of immune reconstitution, engraftment, and donor chimerism resulting from this combined preparative regimen.

III. To determine rates of disease relapse, acute graft-versus-host disease (GVHD), and day 100 disease-free survival in patients receiving 131 I-BC8 antibody (Ab) combined with CY, FLU, 2 Gy TBI, tacrolimus, MMF, and human leukocyte antigen (HLA)-haploidentical allogeneic hematopoietic cell transplant (HCT).

OUTLINE: This is a dose-escalation study of iodine I 131 monoclonal antibody BC8.

RADIOIMMUNOTHERAPY: Patients receive therapeutic iodine I 131 monoclonal antibody BC8 via central line on day -14.

NONMYELOABLATIVE CONDITIONING: Patients receive FLU intravenously (IV) over 30 minutes on days -6 to -2 and CY IV over 1 hour on days -6 and -5. Patients undergo TBI on day -1.

TRANSPLANTATION: Patients undergo allogeneic bone marrow transplantation on day 0.

POST-TRANSPLATATION IMMUNOSUPPRESSION: Patients receive CY IV over 1-2 hours on day 3, MMF IV or orally (PO) thrice daily (TID) on days 4 to 35, and tacrolimus IV over 1-2 hours or PO on days 4 to 180 with taper on day 84.

Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 6, 9, 12, 18, and 24 months, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced AML or ALL defined as beyond first remission, primary refractory disease, or evolved from myelodysplastic or myeloproliferative syndromes; or patients with MDS expressed as refractory anemia with excess blasts (RAEB), refractory cytopenia with multilineage dysplasia (RCMD), RCMD with ringed sideroblasts (RCMD-RS), or chronic myelomonocytic leukemia (CMML)
* Patients not in remission must have cluster of differentiation (CD)45-expressing leukemic blasts; patients in remission do not require phenotyping and may have leukemia previously documented to be CD45 negative (because in remission patients, virtually all antibody binding is to non-malignant cells which make up >= 95% of nucleated cells in the marrow)
* Patients should have a circulating blast count of less than 10,000/mm^3 (control with hydroxyurea or similar agent is allowed)
* Patients must have a creatinine clearance greater than 50/ml per minute by the following formula (test must be performed within 28 days prior to registration):

  * Creatinine clearance (CrCl) = (140-age) (Wt in Kg) x 0.85 (female) OR 1.0 (male)/72 x serum Cr
* Bilirubin < 2 times the upper limit of normal
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2 times the upper limit of normal
* Karnofsky score >= 70 or Eastern Cooperative Oncology Group (ECOG) =< 2
* Patients must have an expected survival of > 60 days and must be free of active infection
* Patients must have a related donor who is identical for one human leukocyte antigen (HLA) haplotype and mismatched at the HLA-A, -B or class II, DR beta 1 (DRB1) loci of the unshared haplotype with the exception of single HLA-A, -B or DRB1 mismatches
* DONOR: Related donor who is identical for one HLA haplotype and mismatched at the HLA-A, -B, or DRB1 loci of the unshared haplotype with the exception of single HLA-A, -B, or DRB1 mismatches

Exclusion Criteria:

* Circulating antibody against mouse immunoglobulin (HAMA)
* Prior radiation to maximally tolerated levels to any critical normal organ
* Cross-match positive with donor
* Patients may not have symptomatic coronary artery disease and may not be on cardiac medications for anti-arrhythmic or inotropic effects
* Left ventricular ejection fraction < 35%
* Corrected diffusion capacity of carbon monoxide (DLCO) < 35% and/or receiving supplemental continuous oxygen
* Liver abnormalities: fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction as evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis, or symptomatic biliary disease
* Patients who are known seropositive for human immunodeficiency virus (HIV)
* Perceived inability to tolerate diagnostic or therapeutic procedures, particularly treatment in radiation isolation
* Central nervous system (CNS) involvement with disease refractory to intrathecal chemotherapy and/or standard cranial-spinal radiotherapy
* Women of childbearing potential who are pregnant (beta-human chorionic gonadotropin positive [b-HCG+]) or breast feeding
* Fertile men and women unwilling to use contraceptives during and for 12 months post-transplant
* Inability to understand or give an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-10-05 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnnie Orozco, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Orozco JJ, Vo PT, Gooley TA, Haaf RL, Lundberg SJ, Hamlin DK, Wilbur DS, Matesan MC, Fisher DR, Gopal AK, Green DJ, Pagel JM, Sandmaier BM. Targeted Radiation Delivery before Haploidentical HCT for High-risk Leukemia or MDS Patients Yields Long-term Survivors. Clin Cancer Res. 2024 Jan 17;30(2):274-282. doi: 10.1158/1078-0432.CCR-23-1200. PMID 37939122

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-six patients enrolled in the study:
  25 - received & completed study treatment
  01 - withdrew because drug preparations failed to meet release criteria for treatment
Pre-assignment Details: Dose escalation plan: single patients will be entered on the first stage, and escalation by 2 Gy increments in the radiation dose delivered to the normal organ receiving the highest dose will occur until a patient experiences a Grade III/IV regimen-related toxicity (Bearman) or dose-limiting toxicity (DLT), at which point the second stage will begin at the next lower dose level. If the first patient (i.e., at the starting dose level) has DLT, de-escalation will occur in 2 Gy increments
Groups:
- Dose Level 1: 12 Gy Iodine-131 + BC8 Monoclonal Antibody; Dose Level 2: 14 Gy Iodine-131 + BC8 Monoclonal Antibody; Dose Level 3: 16 Gy Iodine-131 + BC8 Monoclonal Antibody; Dose Level 4: 18 Gy Iodine-131 + BC8 Monoclonal Antibody; Dose Level 5: 20 Gy Iodine-131 + BC8 Monoclonal Antibody; Dose Level 6: 22 Gy Iodine-131 + BC8 Monoclonal Antibody; Dose Level 7: 24 Gy Iodine-131 + BC8 Monoclonal Antibody; Dose Level 8: 26 Gy Iodine-131 + BC8 Monoclonal Antibody: RADIOIMMUNOTHERAPY: Patients receive therapeutic iodine I 131 monoclonal antibody BC8 via central line on day -14.
  NONMYELOABLATIVE CONDITIONING: Patients receive FLU IV over 30 minutes on days -6 to -2 and CY IV over 1 hour on days -6 and -5. Patients undergo TBI on day -1.
  TRANSPLANTATION: Patients undergo allogeneic bone marrow transplantation on day 0.
  POST-TRANSPLATATION IMMUNOSUPPRESSION: Patients receive CY IV over 1-2 hours on day 3, MMF IV or PO TID on days 4 to 35, and tacrolimus IV over 1-2 hours or PO on days 4 to 180 with taper on day 84.
  Allogeneic Bone Marrow Transplantation: Given via central line
  Cyclophosphamide: Given IV
  Fludarabine Phosphate: Given IV
  Iodine I 131 Monoclonal Antibody BC8: Given IV (dosimetry dose) or via central line (therapeutic dose)
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given IV or PO
  Tacrolimus: Given IV or PO
  Total-Body Irradiation: Undergo TBI
Period: Overall Study
Arm/Group | Dose Level 1: 12 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 2: 14 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 3: 16 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 4: 18 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 5: 20 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 6: 22 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 7: 24 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 8: 26 Gy Iodine-131 + BC8 Monoclonal Antibody
Started | 1 | 1 | 5 | 1 | 1 | 2 | 7 | 7
Completed | 1 | 1 | 5 | 1 | 1 | 2 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: 12 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 2: 14 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 3: 16 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 4: 18 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 5: 20 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 6: 22 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 7: 24 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 8: 26 Gy Iodine-131 + BC8 Monoclonal Antibody | Total
Number analyzed (Participants) | 1 | 1 | 5 | 1 | 1 | 2 | 7 | 7 | 25
Age, Categorical [Count of Participants; unit: Participants] — Population: This is a dose-escalation study.
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 1 | 1 | 5 | 1 | 1 | 2 | 6 | 5 | 22
    >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 3 | 9
  Male | 1 | 1 | 3 | 0 | 0 | 2 | 5 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 1 | 1 | 4 | 1 | 1 | 2 | 7 | 7 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 4
  White | 1 | 0 | 3 | 0 | 1 | 0 | 5 | 5 | 15
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 5 | 1 | 1 | 2 | 7 | 7 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLT) 30 Days After Transplant
Description: The criteria of Grade III/IV regimen-related toxicity (Bearman) or dose-limiting toxicity (DLT) are as follows:
  Grade 1 Development of transient chemical abnormalities which are not of major clinical consequence and which reverse without requiring major medical interventions. In general, the intent of this toxicity scale is to observe transient target organ toxicity which is reversible.
  Grade 2 Development of chemical or laboratory abnormalities that are persistent and which may represent target organ damage that may not be readily reversed. It is anticipated that at this dose of the drug, the toxicity obtained would be manageable by clinical methods but may interfere with other therapies.
  Grade 3 Development of major clinical, chemical or laboratory abnormalities which represent maximum toxicities without being fatal. This grade of toxicity is designed to be the dose-limiting toxicity.
  Grade 4 Fatal
Time Frame: Up to 30 days post-transplant
Population: Number of participants that experienced a dose-limiting toxicity (DLT) within 30 days following transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 12 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 2: 14 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 3: 16 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 4: 18 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 5: 20 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 6: 22 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 7: 24 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 8: 26 Gy Iodine-131 + BC8 Monoclonal Antibody
Number analyzed (Participants) | 1 | 1 | 5 | 1 | 1 | 2 | 6 | 8
Participants
  Number of participants with no dose-limiting toxicities 30 days after transplant | 1 | 1 | 5 | 1 | 1 | 2 | 6 | 7
  Number of participants with dose-limiting toxicities 30 days after transplant | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

2. Secondary Outcome: Number of Participants With Transplant-Related Mortality Within 100 Days After Transplant
Description: Number of Participants that received and completed study treatment who died within 100 days after transplant
Time Frame: Up to 100 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 12 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 2: 14 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 3: 16 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 4: 18 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 5: 20 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 6: 22 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 7: 24 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 8: 26 Gy Iodine-131 + BC8 Monoclonal Antibody
Number analyzed (Participants) | 1 | 1 | 5 | 1 | 1 | 2 | 7 | 7
Participants
  Number of participants who died within 100 days after transplant | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1
  Number of participants who are alive within 100 days after transplant | 1 | 1 | 4 | 1 | 1 | 1 | 5 | 6

3. Secondary Outcome: Participant Disease Response Within 90 Days After Transplant
Description: The number of participants that are in complete remission or relapsed within 90 days after transplant
  Complete Remission is defined as the complete resolution of all signs of leukemia for at least 90 days with all of the following:
  1. Normal bone marrow with blasts <5% with normal cellularity, normal megakarypoiesis, more than 15% erythropoiesis, and more than 25% granulocytopoiesis.
  2. Normalization of blood counts (no blasts, platelets > 100000/mm3, granulocytes >1500/mm3)
  3. No extramedullary disease
  Relapse is measured as follows:
  1. After CR: >5% blasts in the bone marrow and/or peripheral blood. Confirmation of relapse by bone marrow analysis with more than 10% blasts.
  2. After PR: increase of blast cells in the marrow to >50% of those during PR.
  3. Extramedullary disease confirmed cytologically or histologically.
Time Frame: Up to 90 days after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 12 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 2: 14 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 3: 16 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 4: 18 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 5: 20 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 6: 22 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 7: 24 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 8: 26 Gy Iodine-131 + BC8 Monoclonal Antibody
Number analyzed (Participants) | 1 | 1 | 5 | 1 | 1 | 2 | 7 | 7
Participants
  Number of participants that are in complete remission 90 days after transplant | 0 | 1 | 2 | 1 | 1 | 1 | 4 | 3
  Number of participants that relapsed within 90 days after transplant | 1 | 0 | 2 | 0 | 0 | 1 | 3 | 3
  Number of participants with unknown disease response | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

4. Secondary Outcome: Severity of Acute GVHD in Patients Who Completed the Study Treatment
Description: The severity of acute GVHD is measured based on Graft vs Host Disease:
  Grade I +1 to +2 skin rash No gut or liver involvement
  Grade II +3 skin rash or
  * 1 gastrointestinal involvement and/or +1 liver involvement
  Grade III +2 to +4 gastrointestinal involvement and/or
  * 2 to +4 liver involvement with or without a rash
  Grade IV Pattern and severity of GVHD similar to grade 3 with extreme constitutional symptoms or death
Time Frame: 100 days after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 12 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 2: 14 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 3: 16 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 4: 18 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 5: 20 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 6: 22 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 7: 24 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 8: 26 Gy Iodine-131 + BC8 Monoclonal Antibody
Number analyzed (Participants) | 1 | 1 | 5 | 1 | 1 | 2 | 7 | 7
Participants
  Number of participants with Grade 0 - 1 GVHD | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
  Number of participants with Grade 2 GVHD | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 4
  Number of participants with Grade 3 GVHD | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
  Number of participants with unknown GVHD | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1

5. Secondary Outcome: Number of Participants With 100% Donor Chimerism at Day 84
Description: Post-transplant bone marrow and peripheral blood samples were collected on day 84 after transplant for DNA Chimerism Analysis
Time Frame: Day 84 after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 12 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 2: 14 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 3: 16 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 4: 18 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 5: 20 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 6: 22 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 7: 24 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 8: 26 Gy Iodine-131 + BC8 Monoclonal Antibody
Number analyzed (Participants) | 1 | 1 | 5 | 1 | 1 | 2 | 7 | 7
Participants
  100% Donor Chimerism on Day 84 | 1 | 1 | 5 | 0 | 1 | 1 | 4 | 6
  <100% Donor Chimerism on Day 84 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1

6. Secondary Outcome: Two-Year Disease-free Survival of Study Participants Who Completed the Study Regimen
Description: Survival and complete resolution of all signs of leukemia 2 years after transplant with all of the following:
  1, Normal bone marrow with blasts <5% with normal cellularity, normal megakaryopoiesis, more than 15% erythropoiesis, and more than 25% granulocytopoiesis.
  2. Normalization of blood counts (no basts, platelets >100,000/mm3, granulocytes >1,500/mm3) 3. No extramedullary disease.
Time Frame: 2 years post-transplant
Population: Participants who are alive and disease-free 2 years after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 12 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 2: 14 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 3: 16 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 4: 18 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 5: 20 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 6: 22 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 7: 24 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 8: 26 Gy Iodine-131 + BC8 Monoclonal Antibody
Number analyzed (Participants) | 1 | 1 | 5 | 1 | 1 | 2 | 6 | 8
Participants | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Serious adverse events and Other (not including serious adverse events) were monitored and recorded from the time of first exposure to the investigational product (i.e. Iodine 131 + BC8 mAB) through day +100 post-transplant or through patient discharge from the Seattle Cancer Care Alliance (SCCA) system to the patient's primary physician. All-Cause Mortality was monitored/assessed for up to 2 years or through participant survival after completing the study regimen and transplant.
Arm/Group | Dose Level 1: 12 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 2: 14 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 3: 16 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 4: 18 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 5: 20 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 6: 22 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 7: 24 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 8: 26 Gy Iodine-131 + BC8 Monoclonal Antibody
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/1 | 5/5 | 0/1 | 0/1 | 2/2 | 5/7 | 7/7
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 4/5 | 1/1 | 0/1 | 2/2 | 5/7 | 7/7
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 5/5 | 1/1 | 1/1 | 2/2 | 6/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: 12 Gy Iodine-131 + BC8 Monoclonal Antibody (N=1) | Dose Level 2: 14 Gy Iodine-131 + BC8 Monoclonal Antibody (N=1) | Dose Level 3: 16 Gy Iodine-131 + BC8 Monoclonal Antibody (N=5) | Dose Level 4: 18 Gy Iodine-131 + BC8 Monoclonal Antibody (N=1) | Dose Level 5: 20 Gy Iodine-131 + BC8 Monoclonal Antibody (N=1) | Dose Level 6: 22 Gy Iodine-131 + BC8 Monoclonal Antibody (N=2) | Dose Level 7: 24 Gy Iodine-131 + BC8 Monoclonal Antibody (N=7) | Dose Level 8: 26 Gy Iodine-131 + BC8 Monoclonal Antibody (N=7)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asystole (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular Arrythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin GVHD (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — GI GVHD
Mucositis/stomatitis (clinical exam) Anus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis/stomatitis (clinical exam) Oral cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, GU Bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, GU Urethra (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Splenic Hemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Splenic Hemorrhage
Diffuse Alveolar Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GI Bleed (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hepatobiliary/Pancreas - Other (Specify, Liver) (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Liver GVHD
CMV Reactivation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CMV Gastritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Infection - Other (Specify, Blood) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Gram Negative Blood Infection
Infection - Other (Specify, Salivary gland) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with grade 3 or 4 neutrophils (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Infection (Pneumonia) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils Blood (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Coag Negative Staph Infection
Infection with normal ANC or Grade 1 or 2 neutrophils Blood (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Multi Organism Infection
Infection with normal ANC or Grade 1 or 2 neutrophils Blood (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Septic Shock
Infection with normal ANC or Grade 1 or 2 neutrophils Blood (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Pneumonia
Infection with normal ANC or Grade 1 or 2 neutrophils Blood (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Parainfluenza
Infection with normal ANC or Grade 1 or 2 neutrophils Blood (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Lung Infection
Infection with normal ANC or Grade 1 or 2 neutrophils Blood (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Coronavirus
CMV Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Altered Mental Status (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 1 (1)
CNS cerebrovascular ischemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: 12 Gy Iodine-131 + BC8 Monoclonal Antibody (N=1) | Dose Level 2: 14 Gy Iodine-131 + BC8 Monoclonal Antibody (N=1) | Dose Level 3: 16 Gy Iodine-131 + BC8 Monoclonal Antibody (N=5) | Dose Level 4: 18 Gy Iodine-131 + BC8 Monoclonal Antibody (N=1) | Dose Level 5: 20 Gy Iodine-131 + BC8 Monoclonal Antibody (N=1) | Dose Level 6: 22 Gy Iodine-131 + BC8 Monoclonal Antibody (N=2) | Dose Level 7: 24 Gy Iodine-131 + BC8 Monoclonal Antibody (N=7) | Dose Level 8: 26 Gy Iodine-131 + BC8 Monoclonal Antibody (N=7)
Allergic Reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Allergic Reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Chest Tightness
Allergic Reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Face Rash
Allergic Reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Fever
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Platelets decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
WBC decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fluid Overload (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills/Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 7 (7)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Insomnia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Rigors (General disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Erythema of the penis
Excoriation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Skin breakdown/decubitus ulcer
Left Eyelid Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulva cellulitis/irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal Fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 7 (7)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 6 (6) | 7 (7)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dysgeusia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 5 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 6 (6) | 7 (7)
Tongue Sores (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Ecchymosis (HEMORRHAGE/BLEEDING) (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (HEMORRHAGE/BLEEDING) (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 5 (5)
Hematuria (HEMORRHAGE/BLEEDING) (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hemorrhage (Bleeding) (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage-Surgery Site (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage-Retina (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage-Vaginal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage-Left Eye (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage-Petechaie (General disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage-Vaginal Spotting (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspergillus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
BK Virus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
C. Difficile (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CMV Enteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CMV Reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Coag Negative Staph (Infections and infestations) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Enterobacter cloacae (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Enterobacter faecalis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Enterococcus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia coli (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Lactobacillus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polymicrobial Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Strep. Viridans (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Vanco. Resistant Enterococcus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parainfluenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Proteus Mirabalis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rothia Mucilaginosa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RSV (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Edema - Face (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema - Hand (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema - Limb (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Edema - Right Eye (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema - Trunk/Genital (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Volume Overload (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Steroid Induced Diabetes (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bell's Palsy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left Foot Drop (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive Disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Delerium (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Feet Numbness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Blurry Vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain - Abdomen (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) — Splenic pain
Pain - Abdomen (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Pain - Chest (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pain - Urethra (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pain - Headache (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 5 (5) | 4 (4)
Pain - Jaw (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Joint Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pain - Leg (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain - Muscle (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pain - Back (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain - Limb (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain - Hip (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain - Neck (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain - Bones (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain - Cardiac (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain - Head/Neck (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain - Rectal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain - Shoulder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain - Sore Throat (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Nodules (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower Extremity DVT (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fluid Overload (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study accrual has been lower (i.e., 26 total) than the planned target accrual of 50 due to the prioritization of other clinical trials using an alternative radiometal (yttrium-90 [90Y]) and antibody construct (BC8-DOTA).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT00589316/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT00589316/SAP_001.pdf